CLINICAL TRIAL: NCT00668993
Title: The Emotional Freedom Technique (EFT) Versus a Waitlist for Food Cravings: A Randomized Clinical Trial
Brief Title: Randomized Clinical Trial Investigating Efficacy of EFT (Emotional Freedom Technique) for Food Cravings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soul Medicine Institute (Other)
Collaborators: Griffith University (Other)
Responsible Party: Dr Peta Stapleton, Griffith University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SMI-GU-42708
Record Dates: First submitted 2008-04-27; First posted 2008-04-29 (Estimated); Last update posted 2009-09-22 (Estimated); Status verified 2009-09

CONDITIONS: Food Cravings

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- A, B (Experimental): A is treatment group B is waitlist group
  Interventions: Behavioral: EFT - the Emotional Freedom technique

INTERVENTIONS:
Behavioral: EFT - the Emotional Freedom technique — EFT combines cognitive strategies with somatic procedures adapted from acupuncture and related systems for altering the cognitive, behavioural, and neurochemical foundations of psychological problems. It is often referred to as "psychological acupuncture". Few adequately controlled studies have been conducted on EFT however acupuncture has been quite extensively studied, with hundreds of research reports published
  Other Names: EFT is often described as "psychological acupuncture"

SUMMARY:
This pilot study will examine one issue only in weight loss - food cravings in overweight (i.e. BMI between 25-29.9) or obese (BMI greater than 30) consumers. Food craving is hypothesized to be an important intervening causal variable and the development of obesity.

This randomized clinical trial will explore whether a relatively under researched energy based therapeutic procedure, Emotional Freedom Techniques (EFT), can reduce food cravings in participants under laboratory-controlled conditions, and compare this to a waitlist group. The following foods will be tested: chocolate, salty foods (e.g. chips, crisps, salted nuts), sweet carbohydrate foods (eg. cakes, biscuits, soft/soda drinks), carbohydrate foods which are neither sweet nor salty such as white refined foods such as bread), and caffeinated items.

Research examining energy based procedures (e.g. EFT) combines cognitive strategies with somatic procedures adapted from acupuncture and related systems for altering the cognitive, behavioural, and neurochemical foundations of psychological problems. It is often referred to as "psychological acupuncture". Few adequately controlled studies have been conducted on EFT however acupuncture has been quite extensively studied, with hundreds of research reports published (see attached references).

Screening will occur over the telephone with one of the chosen self report questionnaires - the Food Craving Inventory (FCI; White et al., 2002). The FCI is a reliable and valid measure for the assessment of cravings for specific types of foods: High Fats, Sweets, Carbohydrates/Starches, and Fast Food Fats, all of which comprise the higher order construct of "food craving" or the FCI Total score (White et al., 2002). Higher numbers for each of the subscales reflect greater cravings for that food type with the highest score being 185. Scores of 93 or higher during the screen will be used to admit subjects to the next diagnostic interview phase of the trial. In addition, subjects will be asked their weight and height in order to ascertain their BMI and this will be confirmed in the diagnostic interview with a standardized weight machine.

The Structured Clinical Interview (SCID-II; Spitzer, Williams, Gibbon, & First, 1990) has 12 groups of questions corresponding to12 personality disorders and will be used as a diagnostic tool in a face-to-face interview with subjects who are suitable from the telephone screen. The aim is to exclude any active diagnoses from the DSM-IV in order to obtain the purest non clinic sample possible. All subjects will be notified by letter of the outcome of their diagnostic interview and those unsuitable for the trial will be told they did not meet selection criteria. Suitable practitioners who would be able to provide individual support for the food cravings will be provided in written format. Subjects who meet a diagnostic category will be informed of this and appropriate referral will be offered.

Participants will be randomly assigned (using the NHMRC Clinical Trials Centre service) to a free group EFT treatment condition or a non treatment waitlist control condition of the same duration (4 weeks). This design ensures that potential treatment gains are neither due to the mere passage of time nor regression to the mean. To limit attrition from waitlist conditions, several contacts will be made with the waiting clients. Prescheduled phone contacts, for example, may maintain adherence to the waitlist condition.

Prior to treatment all subjects will be weighed and height measured for their BMI status and food craving outcome measures (pre, post and follow-up) will be measured using:

1. SUDS rating (subjective) in daily food diaries (food diaries were chosen as a method that best measures real-life eating behaviour)
2. Power of Food Scale (Didie, 2003)
3. Food Craving Inventory (White et al., 2002)

Three aspects of eating behaviour will be measured using the Revised Restraint Scale (Herman & Polivy, 1980). The items are summed for a total score that ranges from 0 to 40. High scores indicate chronic dieting in which the individual is constantly cycling on and off the diet, typically without any substantial weight loss. Dietary restraint appears to play a causal role in the development of eating disorders and obesity and loss of control over intake. Food cravings may trigger these eating behaviours.

The Symptom Assessment 45 (SA-45, Strategic Advantage, 1998) will be used to assess symptomatology across nine psychiatric domains and as measures of the outcome of the psychological intervention.

Demographic information will be collected in questionnaire format at the beginning of the study.

The EFT intervention will consist of 4 sessions (2 hours duration) with homework and will be based on standard delivery of EFT, as per founder Gary Craig's training for level 1 EFT certification ( see http://www.emofree.com/WorkShop/workshop-guidelines.htm#Level%201).

DETAILED DESCRIPTION:
Participants will be recruited through community announcements in print advertisements, radio, and television. Inclusion and exclusion criteria will be highlighted in the advertising. Criteria will consist of: participants being (l) over 18 years old and under 60 years and not suffering any severe psychological impairment, (2) not currently receiving treatment (psychological or medical) for their food cravings, (3) agree to be contacted for follow-up testing. Women and men will be included, and (4) active diagnoses from the SCID II and subjects taking 'heavy' psychotropic (see attached list) which can suppress feelings, cravings and sensitivity will be excluded.

Known sufferers of diabetes (Type I and II) and hypoglycemia will be excluded due to any physiological aetiology (effects related) to food cravings.

Eligible applicants will be offered participation in the study through an informed consent procedure. Self report questionnaires will be issued as part of the study and a demographic questionnaire will be included in this. All identifying information will be destroyed once data has been analysed.

Unsuitable participants will be advised in letter form that they did not meet selection criteria, and a list of suitable practitioners will be included should they wish to address their food craving.The study will use a Research Assistant to screen participants, administer questionnaires and collate data. Separate qualified clinicians to the investigating researchers will be used to deliver the EFT treatment condition.

The treatments will be delivered in a number of appropriate venues. Analysis will examine pre versus post effects for each intervention to highlight any differences in self report, and a repeated measures ANOVA will examine the effect of time on all the self report scores.

The following questions will be addressed: does EFT reduce food cravings and weight more than no intervention? It is anticipated that because this is a pilot study, results may indicate positive direction for these questions only. Due to anecdotal suggestion that EFT has long lasting effects (see http://www.emofree.com/articles.aspx?id=19), it is hypothesised that food cravings will reduce significantly with the EFT intervention and remain consistent at follow-up points. It is expected that the waitlist condition will remain unaffected prior to any treatment condition. Increases in eating restraint and decreases in SUDS ratings and general psychopathology are expected with the EFT intervention post treatment and are expected to stay constant at 3-, 6- and 12-month follow-up. Gender and age will be examined.

A standard process will be used for informed consent, including a general information sheet for subjects and consent form indicating any areas of psychological risk, benefits of the study, self report questionnaire details and follow-up procedures. Detailed information about what constitutes a food craving will be given to all subjects as well as information about voluntary involvement and study withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Criteria will consist of participants being:

  l) over 18 years old and under 60 years and not suffering any severe psychological impairment

  2) not currently receiving treatment (psychological or medical) for their food cravings

  3) agree to be contacted for follow-up testing.
* Women and men will be included

Exclusion Criteria:

* Active diagnoses from the SCID II and subjects taking 'heavy' psychotropic which can suppress feelings, cravings and sensitivity will be excluded.
* Known sufferers of diabetes (Type I and II) and hypoglycemia will be excluded due to any physiological aetiology (effects related) to food cravings.
* Pregnant women will be excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Decrease or elimination of food craving | 6 and 12 months follow up

SECONDARY OUTCOMES:
changes in weight | 6 and 12 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Peta Stapleton, PhD, Principal Investigator — Griffith University
Locations (1):
- School of Medicine, Meadowbrook, Queensland, Australia